CLINICAL TRIAL: NCT01907568
Title: Understanding Hallucinations (Part I) - Phenomenology and Cognition
Brief Title: Understanding Hallucinations (Part I)
Acronym: UH-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: University Medical Center Groningen (Other); Free University Medical Center (Other); Parnassia Groep (Other)
Responsible Party: Principal Investigator, Iris Sommer, Prof.Dr., UMC Utrecht
Other Study IDs: UH-1; NL42959.041.13 (Other: Toetsingonline)
Record Dates: First submitted 2013-07-08; First posted 2013-07-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Hallucinations; No Hallucinations
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (11):
- Patients with schizophrenia: With and without hallucinations
- Patients with borderline personality disorder: With and without hallucinations
- Patients with hearing impairment: With and without hallucinations
- Patients with visual loss: With and without hallucinations
- Patients with Parkinson's Disease: With and without hallucinations
- Patients with Alzheimer's Disease: With and without hallucinations
- Patients with dementia with Lewy Bodies: With and without hallucinations
- Patients with Posttraumatic Stress Disorder: With and without hallucinations
- Patients with delirium: With and without hallucinations
- Healthy participants: With and without hallucinations
- Patients with mood disorder: With and without hallucinations

SUMMARY:
Psychotic symptoms (hallucinations and delusions) are present in several psychiatric and neurological disorders as well as in the general population. Effective treatment strategies for these symptoms in all patients are lacking and treatment-response can presently not be predicted. To date, the exact pathophysiological mechanism of these symptoms remains unknown. By investigating (subtypes) of hallucinations and delusions in all populations, a common pathway may be found, leading to more effective treatment options. Alternatively, different subtypes may be associated with different pathophysiological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* mentally competent
* in case of delirium: family member able to give informed consent
* Individuals with hallucinations will have to experience at least one episode of hallucinations over the last month.
* Individuals without hallucinations: no current hallucinations and a history of maximum 1 episode of hallucinations with a maximum duration of 1 week, at least two years ago.

Exclusion Criteria:

* Age <18)
* Participants that cannot read, speak or understand Dutch
* For all included diagnostic groups except delirium: Mentally incompetent individuals who are not capable to provide informed consent, as determined by their treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to include subjects of each of the following diagnostic groups, both with and without psychotic symptoms:
  1. patients with schizophrenia spectrum disorders
  2. patients with borderline personality disorder (BPD)
  3. patients with hearing impairment
  4. patients with visual loss
  5. patients with Parkinson's disease (PD)
  6. patients with Alzheimer's disease (AD)
  7. patients with Lewy Body dementia (DLB)
  8. patients with post-traumatic stress disorder (PTSD)
  9. patients with delirium
  10. healthy individuals
  11. patients with mood disorder
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The number of clusters of patients with shared symptom profiles as determined by latent class analysis, and the difference in scores on cognitive assessment between these identified clusters. | Three years

SECONDARY OUTCOMES:
The internal consistency, test-retest reliability, inter-rater reliability, criterion validity and construct validity of a newly developed questionnaire. | Two years
The difference in scores on cognitive assessment between participant groups with and without psychotic symptoms. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, Prof, MD, PhD, Principal Investigator — UMC Utrecht; Teus van Laar, MD, PhD, Principal Investigator — UMC Groningen; Philip Scheltens, Prof, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Karin Slotema, MD, PhD, Principal Investigator — Parnassia Groep
Locations (4):
- Netherlands (4):
  - VU Medical Center, Amsterdam
  - UMC Groningen, Groningen
  - Parnassia Bavo Groep, The Hague
  - UMC Utrecht, Utrecht